CLINICAL TRIAL: NCT00602199
Title: A Phase II Study of Anti-angiogenesis Therapy for Metastatic Melanoma Using ABT-510
Brief Title: ABT-510 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Svetomir Nenad Markovic, M.D., Mayo Clinic
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000582475; P30CA015083 (NIH); MC0375 (Other: Mayo Clinic Cancer Center); 1439-04 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-01-11; First posted 2008-01-28 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma
MeSH Terms: conditions — Melanoma | interventions — NAc-Sar-Gly-Val-(d-allo-Ile)-Thr-Nva-Ile-Arg-ProNEt; Immunoenzyme Techniques; Immunohistochemistry; Biopsy

INTERVENTIONS:
Drug: ABT-510
Other: immunoenzyme technique
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Other: pharmacological study
Procedure: biopsy

SUMMARY:
RATIONALE: ABT-510 may stop the growth of melanoma by blocking blood flow to the tumor.

PURPOSE: This phase II trial is studying how well giving ABT-510 works in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Examine the safety profile of ABT-510 in patients with metastatic malignant melanoma.
* Examine the antitumor activity (i.e., time to progression and response rates) in patients treated with ABT-510.
* Determine the pharmacodynamic effects of ABT-510 and its potential impact on immune cell function in these patients.

OUTLINE: Patients receive ABT-510 subcutaneously twice daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

Blood samples are obtained at baseline, before treatment on day 1 of cycles 2 and 3, and then every other course thereafter for pharmacological and ancillary studies. Samples are evaluated for EC enumeration, expression profiling, circulating tumor cell quantification, analysis of T-cell functions (i.e., immunophenotyping for NK-, T- and B-cell phenotypes as well as ELISPOT analysis against common environmental pathogens and T cell spectratyping), and angiogenesis bioassays. Patients also undergo ultrasound-guided core tumor biopsies for histological analysis of microvascular density (CD38 and von Willebrand Factor immunohistochemistry) at baseline and before treatment on day 1 of courses 3 and 5.

After completion of study treatment, patients are followed every 3 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed malignant melanoma

  * Stage IV disease
  * No known potentially curative standard therapy that exists or is proven capable of extending life expectancy
* Measurable disease
* No history of or current CNS metastases

  * MRI of the brain to confirm absence of CNS metastases within the past 28 days is required
* No known, presently active carcinomatous meningitis

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 6 months
* ANC ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Alkaline phosphatase ≤ 3 times upper limit of normal (ULN)
* AST ≤ 3 times ULN
* Creatinine ≤ 2.5 times ULN
* Hemoglobin ≥ 9.0 g/dL
* Prothrombin time normal
* Willing to return to Mayo Clinic Rochester, Jacksonville or Scottsdale for follow-up
* Must be able to self-administer or has a caregiver who can reliably administer subcutaneous injections
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No uncontrolled or current infection
* No New York Heart Association class III-IV heart disease
* No recent history of (i.e., ≤ 12 weeks from study day 1) or current cancer-related bleeding event (e.g., hemoptysis)
* No recent history of (within the past 4 weeks) or current noncancer-related clinically significant bleeding event
* No uncontrolled hypertension
* No history of stroke or other CNS bleeding events (e.g., aneurysms)

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior chemotherapy and recovered (6 weeks for mitomycin C or nitrosoureas)
* At least 4 weeks since prior immunotherapy, biologic therapy, radiotherapy, or surgery
* No concurrent anticoagulation therapy or antiplatelet therapy
* No other concurrent antineoplastic agents (e.g., cytotoxic chemotherapy, immunotherapy, radiotherapy, or investigational therapy) except local radiotherapy for supportive reasons involving a small radiation field

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2004-11; Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

PRIMARY OUTCOMES:
18-week progression-free survival rate

SECONDARY OUTCOMES:
Objective response rate as defined by RECIST criteria
Overall survival time
Frequency of NK-cells, T-cells, and B-cells before the start of the first 5 courses of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Svetomir Markovic, MD, PhD, Study Chair — Mayo Clinic

REFERENCES:
- [Result] Markovic SN, Suman VJ, Rao RA, Ingle JN, Kaur JS, Erickson LA, Pitot HC, Croghan GA, McWilliams RR, Merchan J, Kottschade LA, Nevala WK, Uhl CB, Allred J, Creagan ET. A phase II study of ABT-510 (thrombospondin-1 analog) for the treatment of metastatic melanoma. Am J Clin Oncol. 2007 Jun;30(3):303-9. doi: 10.1097/01.coc.0000256104.80089.35. PMID 17551310